CLINICAL TRIAL: NCT04627350
Title: Early Detection of Lung Cancer in Czech High-risk Asymptomatic Individuals
Acronym: ELEGANCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Lukas Lambert, Associated professor, General University Hospital, Prague
Other Study IDs: R01
Record Dates: First submitted 2020-08-27; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Lung Cancer
Keywords: lung cancer; low dose CT
MeSH Terms: conditions — Lung Neoplasms | interventions — Fibrillins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LDCT: Single arm - all patients undergo low-dose CT (LDCT) examination of lungs
  Interventions: Other: Response to pulmonary finding (nodule, mass)

INTERVENTIONS:
Other: Response to pulmonary finding (nodule, mass) — Follow-up low-dose CT, PET-CT, tissue sampling (transparietal biopsy, bronchoscopy, resection), contrast-enhanced CT of the thorax

SUMMARY:
The aim of this study is to evaluate and optimize entry criteria for the proposed programme for early detection of lung cancer in the Czech Republic.

An estimated 3200 high-risk (age 55-74 years, >30 pack-years) asymptomatic individuals will undergo baseline low-dose chest CT (LDCT) and a follow-up LDCT at 1 year. Patients with poor performance status (PS) 2-4, history of malignancy in the past 10 years, chest CT in the past 1 year, bodyweight >140kg will not be included.

The patients will fill out a questionnaire with basic data, including smoking history (pack-years), history of previous malignancy, CT imaging of the thorax, and will undergo spirometry.

Outcomes of the study include:

* optimization of entry criteria, optimization of timing of a follow-up LDCT and management of the patients, proposal of quality assurance indicators
* influence of screening on the stage of lung cancer at the time of the diagnosis and life-years lost
* cost-effectiveness of the screening program
* evaluation of the diagnostic yield for secondary findings (pulmonary fibrosis, cardiovascular risk)

ELIGIBILITY:
Inclusion Criteria:

* Age 55-74 years
* Smoking: >= 30 pack-years, smoker or ex-smoker <15 years
* Performance status (0-1) - can climb at least one floor without any difficulty or pause

Exclusion Criteria:

* Body weight above 140 kg
* Malignant disease within the last 10 years (except non-melanoma skin cancer).
* Chest CT less than one year ago
* Clinical signs suspicious of lung cancer (weight loss, new cough, hemoptysis)

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Defined by eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of cancers detected at stage I | 2023
  The proportion of cancers diagnosed at a resectable stage (stage I) vs. non-resectable stage (II-IV) will be compared to the stage distribution in an unscreened population

SECONDARY OUTCOMES:
The cost per diagnosis at a resectable stage | 2023
  The cost per diagnosis at a resectable stage will encompass the cost of low-dose CT (LDCT), follow-up LDCT, verification (PET/CT, tissue sampling, bronchoscopy).

OTHER OUTCOMES:
Number of secondary examinations | 2023
  The number, cost, and complications of secondary examinations generated by screening LDCT.
Number of secondary findings | 2023
  The number and types of secondary findings and their clinical relevance (potentially important vs. unimportant findings) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Lambert, M.D., Principal Investigator — General University Hospital, Prague
Locations (1):
- General University Hospital in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.